CLINICAL TRIAL: NCT00156130
Title: Accelerated Radiotherapy Outcomes in Women (Long Term Outcomes of a Randomized Trial of Breast Irradiation Schedules After Lumpectomy in Women With Node-Negative Breast Cancer)(AROW)
Brief Title: Accelerated Radiotherapy Outcomes in Women
Status: Completed | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: OCOG-2003-AROW; CBCRI-Grant-014366
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Lumpectomy; Radiotherapy; Hypofractionated Radiotherapy; Long Term Outcomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Accelerated whole breast irradiation
  Interventions: Radiation: Accelarated radiotherapy schedule
- 2: Conventional whole breast irradiation
  Interventions: Radiation: Conventional radiotherapy schedule

INTERVENTIONS:
Radiation: Conventional radiotherapy schedule — 50 Gy in 25 fractions over 35 days
  Groups: 2
Radiation: Accelarated radiotherapy schedule — 42.5 Gy in 16 fractions over 22 days
  Groups: 1

SUMMARY:
This study is evaluating the long-term outcomes of women in a randomized trial that compared accelerated whole breast irradiation (42.5 Gy in 16 fractions over 22 days) to a longer conventional schedule of whole breast irradiation (50 Gy in 25 fractions over 35 days) following breast-conserving surgery. The outcomes evaluated will include cosmetic outcome and cardiac disease as a measure of late radiation morbidity and local breast recurrence as a measure of effectiveness.

DETAILED DESCRIPTION:
This study is evaluating the long-term outcomes of women in a randomized trial that compared accelerated whole breast irradiation (42.5 Gy in 16 fractions over 22 days) to a longer conventional schedule of whole breast irradiation (50 Gy in 25 fractions over 35 days) following breast-conserving surgery. The results reported at 5 years demonstrated equivalence for these two different radiation schedules for the effect of local recurrence in the breast and cosmetic outcome. Emerging data has suggested that accelerated or shorter radiation schedules may potentially be associated with an increased risk of late morbidity of the skin, soft tissue and the heart at 10 years and beyond. The purpose of this study is to evaluate the long term outcomes of women randomized in the trial. The outcomes evaluated will include cosmetic outcome and cardiac disease as a measure of late radiation morbidity and local breast recurrence as a measure of effectiveness.

ELIGIBILITY:
Only patients recruited into the "Randomized Trial of Hypofractionated Radiotherapy Post-Lumpectomy in Women with Node Negative Breast Cancer" study are eligible to be enrolled into this study.

Inclusion Criteria:

1. The female patient has a histological diagnosis of invasive carcinoma of the breast, and no evidence of metastatic disease.
2. Has had a lumpectomy (including segmental resection and partial mastectomy), that is, surgical excision of the tumour with a rim of normal tissue.
3. Patient has not had an axillary dissection, OR for patients who have had an axillary dissection, all nodes are negative for metastatic disease.

Exclusion Criteria:

1. Tumour greater than 5 cm in greatest diameter on pathological examination.
2. The presence of invasive or intraductal (noninvasive) breast cancer involving the surgical margins.
3. Clinical evidence prior to surgery of infiltration of the skin of the involved breast such as edema, ulceration, or fixation of the tumour to underlying muscle, or inflammatory breast cancer.
4. Bilateral malignancy of the breast (synchronous or metachronous).
5. More than one primary invasive tumour in the same breast.
6. Previous surgery for breast cancer.
7. Pathological status of axilla is unknown.
8. Status for adjuvant systemic therapy not determined.
9. For patients not treated with adjuvant chemotherapy: unable to commence radiation therapy within 16 weeks of last surgical procedure on the breast.
10. For patients treated with adjuvant chemotherapy: unable to commence radiation therapy within 8 weeks of the last dose of chemotherapy.
11. Serious nonmalignant disease (eg. cardiovascular, renal, etc.) which would preclude surgical or radiation treatment.
12. Currently pregnant or lactating.
13. Breast deemed too large to permit satisfactory radiation (ie. separation > 25 cm).
14. Previous concomitant malignancies of any type except squamous, or basal cell carcinomas of the skin, or carcinoma in situ of the cervix which have been effectively treated.
15. Geographic inaccessibility for follow-up.
16. Psychiatric or addictive disorders which preclude obtaining informed consent or adherence to the protocol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extended long term follow-up of patients recruited into the "Randomized Trial of Hypofractionated Radiotherapy Post-Lumpectomy in Women with Node Negative Breast Cancer" study.
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2003-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whelan, MD, Study Chair — Juravinski Cancer Centre
Locations (11):
- Canada (11):
  - Regional Cancer Program of the Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital-Integrated Cancer Program, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Regional Cancer Care - Thunder Bay HSC, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - The Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Montreal General Hospital, Montreal, Quebec